CLINICAL TRIAL: NCT02873715
Title: The Effectiveness of Family-based Weight Loss Treatment Implemented in Primary Care Centers
Brief Title: Primary Care Pediatrics Learning Activity and Nutrition With Families
Acronym: PLAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1131521-174563; U01HL131552 (NIH)
Record Dates: First submitted 2016-08-17; First posted 2016-08-19 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Obesity
Keywords: Childhood weight control
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor will be blinded to the families group assignment. Coaches will be back up assessor. Coach 1 will be an assessor for families assigned to Coach 2, Coach 2 will collect measures for families assigned to Coach 3, and Coach 3 will collect measures for families assigned to Coach 1. Thus, coaches will not collect height and weight measures for families from their caseload.
  Although not possible to guarantee that coaches are blind to condition for families that are not in their caseload due to the families not being blinded, use of a standard protocol (see Appendix C) ensures objective and reliable measurement of the primary outcome. Assessors will be blind to prior heights/weights, further protecting against assessment bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (UC) (Active Comparator): Usual Care will consist of the care typically delivered by the family's primary care provider for children with overweight or obesity. The implementations of UC may vary between providers but typically includes and assessment of the child's weight, help remove barriers to weight loss and introductions of goals for better weight management.
  Interventions: Behavioral: Usual Care
- Family-based treatment (FBT) (Experimental): Family- Based treatment utilizes behavior change techniques to target family-wide changes in diet and physical activity habits with the goal of promoting weight loss and subsequently healthy weight maintenance in all participants. Participants will have visits between 30 to 60 minutes as frequent as weekly and no longer than monthly over the two year study
  Interventions: Behavioral: Family-based treatment; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Family-based treatment — Family based treatment as the invention to randomized participants. Family Based treatment utilizes behavior change techniques to target family-wide changes in diet and physical activity habits with the goal of promoting weight loss and subsequently healthy weight maintenance in all participants. Participants will have visits between 30 to 60 minutes as frequent as weekly and no longer than monthly over the two year study
  Other Names: FBT
  Arms: Family-based treatment (FBT)
Behavioral: Usual Care — Usual care is a treatment that is normally provided to patients in pediatric offices by a pediatrician, physician assistant, or other primary care staff.
  Other Names: UC

SUMMARY:
This study is designed to translate an evidence-based family-based weight loss treatment for childhood obesity (FBT) into primary care settings using co-located interventionists to serve as a model for care delivered within a patient-centered medical home. FBT will be compared to usual care (UC), and the families will be followed for a 2 year period to assess between group differences in the targeted child and parent outcomes, weight changes in non-targeted siblings who are overweight/obese, parent and child changes in delay of gratification, and how these changes relate to weight loss, and the assessment of how provider attitudes predict their intention to use FBT in the future. The results of this study will inform future dissemination and implementation of FBT into primary care settings.

DETAILED DESCRIPTION:
Family-based treatment (FBT) is a behavioral weight control intervention that targets children who have overweight/obesity and their parents, and has the capacity to improve the weight status of non-targeted family members such as siblings. FBT has significant positive effects on body weight in children for up to 10-years of follow-up, and a robust relationship is observed between child and parent outcomes. FBT's concurrent care of two generations of obesity in the family is more efficacious and cost-effective than if family members are treated by their separate health care providers. Despite its recognized efficacy, FBT is mainly available in specialty clinics and many children fail to receive this guideline-based level of treatment, as recommended by the U.S. Preventive Services Task Force. Primary care offers an optimal setting for delivery of FBT by capitalizing on the established relationship between primary care providers and families. Using interventionists co-located within the primary care setting overcomes barriers posed by fragmentation of care, and lack of provider time and training. One of the challenges to integrating childhood obesity treatment into primary care is optimizing limited health care resources. In behavioral weight loss programs, some individuals learn diet, physical activity, and behavior change information quickly, while others learn more slowly. Individuals also differ in their ability to implement treatment recommendations due to individual differences, such as problems with delaying gratification. FBT accommodates these individual differences by using a personalized system of instruction, or a mastery model, in which the content and dose of treatment is calibrated to the needs of the family, ensuring that treatment effort is consistent with need. This multi-site, clinical trial aims to evaluate over a two year period the effectiveness of FBT delivered by a trained interventionist co-located within primary care plus usual care delivered by the primary care provider (FBT) compared to usual care (UC). Participants will be a representative sample of 528 families with a 6-12 year-old child and a parent who have both overweight/obesity. Weight changes in approximately 228 siblings who have overweight/obesity and between 2-18 years of age will also be studied. This study will test between group differences in child (Primary Specific Aim 1A) and parent (Secondary Specific Aim 1) weight change, as well as weight change in siblings who have overweight/obesity (Secondary Aim 2), changes in parent and child delay of gratification, and how changes in delay of gratification are related to parent and child weight changes (Secondary Aim 3), participant level predictors of treatment success (Secondary Aim 4), and how provider attitudes toward evidence-based treatment and perceptions of FBT may relate to their intention to use colocated FBT in their practices in the future (Exploratory Aim 1). Establishing that FBT can be effectively implemented within real world settings is crucial to creating a system by which children and their families who suffer from obesity can be treated in a centralized primary care setting.

ELIGIBILITY:
Inclusion criteria:

The participating child will be between the ages of 6 and 12 and have a BMI above the 85th percentile for age and sex. The participating child will have at least one parent who has overweight or obesity (BMI>25) and who must agree to attend all parent/child treatment meetings as the participating parent. For families in which one parent has overweight/obesity, this parent will be required to be the participating parent in order for the family to be eligible for the study; if two parents have overweight/obesity, the family will choose one parent to enroll in the study. Similarly, if two children in the family have overweight/obesity, it will be encouraged that the older sibling be the primary participant, as it is more likely the younger sibling will model the older sibling. Though only the child who has overweight/obesity and the participating parent will be required to attend treatment sessions, all family members living in the household, including other adults and siblings, will be encouraged to participate indirectly by supporting changes in the family's lifestyle. Because a secondary aim of the study involves the tracking of treatment effects through the household to non-targeted siblings, heights and weights of at least one sibling with overweight/obesity (BMI>85th percentile for age and sex)in the family will be collected, if applicable. Only siblings ages 2- 18 would qualify. All participants must be able to speak and comprehend English at a first-grade level.

Exclusion Criteria:

The participating parent or child will not have had a concussion in the past three months; will not have any significant developmental delays or intellectual disabilities; will not be receiving treatment for a Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-5) disorder that interferes with treatment delivered as part of the intervention; will not have a physical disability or diagnosis that prevents performance of physical activity at a level equivalent to a brisk walk or that places severe restriction on diet; will not be on a medication regimen that affects weight; will not have a medical condition that alters nutritional status, intestinal absorption, or affects weight; will not have undergone weight loss surgery; and will not be participating in an alternate weight control program. Families in which either the participating child or parent is actively involved in other weight-loss treatment, is using weight-affecting medications, or has an impairing psychiatric or medical condition that would hinder participation in the study will be excluded as identified by the screening assessments. Families that are planning to move or in which the participating parent is pregnant or is planning on becoming pregnant during the 2 year study period will also be excluded.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H Epstein, PhD, Principal Investigator — State University of New York at Buffalo; Denise Wilfley, PhD, Principal Investigator — Washington University in Saint Louis; Ken Schechtman, PhD, Principal Investigator — Washington University in Saint Louis
Locations (4):
- United States (4):
  - Washington University in St. Louis, St Louis, Missouri
  - University at Buffalo, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - Nationwide Childrens Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolko RP, Kass AE, Hayes JF, Levine MD, Garbutt JM, Proctor EK, Wilfley DE. Provider Training to Screen and Initiate Evidence-Based Pediatric Obesity Treatment in Routine Practice Settings: A Randomized Pilot Trial. J Pediatr Health Care. 2017 Jan-Feb;31(1):16-28. doi: 10.1016/j.pedhc.2016.01.001. Epub 2016 Feb 9. PMID 26873293
- [Background] Maddison R, Marsh S, Foley L, Epstein LH, Olds T, Dewes O, Heke I, Carter K, Jiang Y, Mhurchu CN. Screen-Time Weight-loss Intervention Targeting Children at Home (SWITCH): a randomized controlled trial. Int J Behav Nutr Phys Act. 2014 Sep 10;11:111. doi: 10.1186/s12966-014-0111-2. PMID 25204320
- [Background] Epstein LH, Paluch RA, Wrotniak BH, Daniel TO, Kilanowski C, Wilfley D, Finkelstein E. Cost-effectiveness of family-based group treatment for child and parental obesity. Child Obes. 2014 Apr;10(2):114-21. doi: 10.1089/chi.2013.0123. Epub 2014 Mar 21. PMID 24655212
- [Background] Quattrin T, Roemmich JN, Paluch R, Yu J, Epstein LH, Ecker MA. Efficacy of family-based weight control program for preschool children in primary care. Pediatrics. 2012 Oct;130(4):660-6. doi: 10.1542/peds.2012-0701. Epub 2012 Sep 17. PMID 22987879
- [Background] Theim KR, Sinton MM, Stein RI, Saelens BE, Thekkedam SC, Welch RR, Epstein LH, Wilfley DE. Preadolescents' and parents' dietary coping efficacy during behavioral family-based weight control treatment. J Youth Adolesc. 2012 Jan;41(1):86-97. doi: 10.1007/s10964-011-9728-5. Epub 2011 Nov 12. PMID 22081241
- [Derived] Button AM, Paluch RA, Schechtman KB, Wilfley DE, Geller N, Quattrin T, Cook SR, Eneli IU, Epstein LH. Parents, but not their children, demonstrate greater delay discounting with resource scarcity. BMC Public Health. 2023 Oct 12;23(1):1983. doi: 10.1186/s12889-023-16832-z. PMID 37828503
- [Derived] Epstein LH, Rizwan A, Paluch RA, Temple JL. Delay Discounting and the Income-Food Insecurity-Obesity Paradox in Mothers. J Obes. 2023 Sep 19;2023:8898498. doi: 10.1155/2023/8898498. eCollection 2023. PMID 37766882
- [Derived] Epstein LH, Wilfley DE, Kilanowski C, Quattrin T, Cook SR, Eneli IU, Geller N, Lew D, Wallendorf M, Dore P, Paluch RA, Schechtman KB. Family-Based Behavioral Treatment for Childhood Obesity Implemented in Pediatric Primary Care: A Randomized Clinical Trial. JAMA. 2023 Jun 13;329(22):1947-1956. doi: 10.1001/jama.2023.8061. PMID 37314275
- See also: Ten-year outcomes of behavioral family-based treatment for childhood obesity. Epstein, Leonard H.; Valoski, Alice; Wing, Rena R.; McCurley, James Health Psychology, Vol 13(5), Sep 1994, 373-383. http://dx.doi.org/10.1037/0278- — https://pubmed.ncbi.nlm.nih.gov/7805631/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each sites local pediatric practices participated in warm hand offs to embeded coaches in the practices to recruit interested families. Families included a targeted child, targeted parent and could include one or multiple siblings but was not required. Recruitment started in November 2017 through August 2019.
Pre-assignment Details: Eligible families were randomized through REDCap directly after completing the screening visit before starting the treatment phase.
Units Other Than Participants: families
Period: Overall Study
Arm/Group | Usual Care (UC) | Family-based Treatment (FBT)
Started | 504; 226 families (226 children and parents, 52 siblings) | 506; 226 families (226 parents and children, 54 siblings)
6-month Follow-up | 403; 199 families (199 children, 164 parents, 40 siblings) | 405; 201 families (201 children, 161 parents, 43 siblings)
12-month Follow-up | 380; 195 families (194 children, 151 parents, 35 siblings) | 386; 199 families (197 children, 148 parents, 41 siblings)
18-month Follow-up | 380; 189 families (189 children, 152 parents, 39 siblings) | 364; 189 families (185 children, 139 parents, 40 siblings)
24-month Follow-up | 413; 205 families (204 children, 172 parents, 37 siblings) | 386; 198 families (196 children, 150 parents, 40 siblings)
Completed | 413; 205 families (204 children, 172 parents, 37 siblings) | 386; 198 families (196 children, 150 parents, 40 siblings)
Not Completed | 91; 21 families | 120; 28 families
Not completed — Lost to Follow-up | 84 | 94
Not completed — Withdrawal by Subject | 7 | 26

BASELINE CHARACTERISTICS:
Population: Parents, targeted children are included in the baseline analysis
Groups:
- Family-based Treatment (FBT): Family- Based treatment utilizes behavior change techniques to target family-wide changes in diet and physical activity habits with the goal of promoting weight loss and subsequently healthy weight maintenance in all participants. Participants will have visits between 30 to 60 minutes as frequent as weekly and no longer than monthly over the two yeart study
  Family-based treatment: Family based treatment as the invention to randomized participants. Family Based treatment utilizes behavior change techniques to target family-wide changes in diet and physical activity habits with the goal of promoting weight loss and subsequently healthy weight maintenance in all participants. Participants will have visits between 30 to 60 minutes as frequent as weekly and no longer than monthly over the two year study
  Usual Care: Usual care is a treatment that is normally provided to patients in pediatric offices by a pediatrician, physician assistant, or other primary care staff.
- Total: Total of all reporting groups
Arm/Group | Usual Care (UC) | Family-based Treatment (FBT) | Total
Number analyzed (Participants) | 504 | 506 | 1010
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The population includes parents, children and siblings which differs between groups and families enrolled.
  years
    Index children: number analyzed (Participants) | 226 | 226 | 452
    Index children | 9.7 (1.9) | 9.8 (1.9) | 9.7 (1.9)
    Parents: number analyzed (Participants) | 226 | 226 | 452
    Parents | 41.4 (7.0) | 41.2 (7.8) | 41.3 (7.5)
    Siblings: number analyzed (Participants) | 52 | 54 | 106
    Siblings | 10.4 (3.8) | 9.7 (3.6) | 10.0 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The total population includes targeted children, parents and siblings. Each row seperately identifies the targeted children, parents and siblings.
  Participants
    Targeted Children: number analyzed (Participants) | 226 | 226 | 452
    Targeted Children: Female | 122 | 120 | 242
    Targeted Children: Male | 104 | 106 | 210
    Parents: number analyzed (Participants) | 226 | 226 | 452
    Parents: Female | 192 | 196 | 388
    Parents: Male | 34 | 30 | 64
    Siblings: number analyzed (Participants) | 52 | 54 | 106
    Siblings: Female | 30 | 30 | 60
    Siblings: Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The total population includes targeted children, parents and siblings. Each row seperately identifies the targeted children, parents and siblings.
  Participants
    Targeted Children: number analyzed (Participants) | 226 | 226 | 452
    Targeted Children: Hispanic or Latino | 19 | 21 | 40
    Targeted Children: Not Hispanic or Latino | 207 | 205 | 412
    Targeted Children: Unknown or Not Reported | 0 | 0 | 0
    Parents: number analyzed (Participants) | 226 | 226 | 452
    Parents: Hispanic or Latino | 8 | 17 | 25
    Parents: Not Hispanic or Latino | 218 | 209 | 427
    Parents: Unknown or Not Reported | 0 | 0 | 0
    Siblings: number analyzed (Participants) | 52 | 54 | 106
    Siblings: Hispanic or Latino | 5 | 6 | 11
    Siblings: Not Hispanic or Latino | 47 | 48 | 95
    Siblings: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The total population includes targeted children, parents and siblings. Each row seperately identifies the targeted children, parents and siblings.
  Participants
    Targeted Children: number analyzed (Participants) | 226 | 226 | 452
    Targeted Children: American Indian or Alaska Native | 1 | 0 | 1
    Targeted Children: Asian | 3 | 5 | 8
    Targeted Children: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Targeted Children: Black or African American | 65 | 58 | 123
    Targeted Children: White | 127 | 131 | 258
    Targeted Children: More than one race | 22 | 17 | 39
    Targeted Children: Unknown or Not Reported | 8 | 15 | 23
    Parents: number analyzed (Participants) | 226 | 226 | 452
    Parents: American Indian or Alaska Native | 0 | 0 | 0
    Parents: Asian | 3 | 3 | 6
    Parents: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parents: Black or African American | 55 | 58 | 113
    Parents: White | 139 | 148 | 287
    Parents: More than one race | 2 | 1 | 3
    Parents: Unknown or Not Reported | 27 | 16 | 43
    Siblings: number analyzed (Participants) | 52 | 54 | 106
    Siblings: American Indian or Alaska Native | 1 | 0 | 1
    Siblings: Asian | 0 | 1 | 1
    Siblings: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Siblings: Black or African American | 13 | 12 | 25
    Siblings: White | 21 | 27 | 48
    Siblings: More than one race | 5 | 5 | 10
    Siblings: Unknown or Not Reported | 12 | 9 | 21
Participants [Count of Participants; unit: Participants]
  Targeted children | 226 | 226 | 452
  Parents | 226 | 226 | 452
  Siblings | 52 | 54 | 106
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. Population: The total population includes targeted children, parents and siblings. Each row seperately identifies the targeted children, parents and siblings.
  kg/m^2
    Targeted Children: number analyzed (Participants) | 226 | 226 | 452
    Targeted Children | 26.9 (5.2) | 26.7 (5.0) | 26.8 (5.1)
    Parents: number analyzed (Participants) | 226 | 226 | 452
    Parents | 37.5 (7.9) | 36.5 (7.6) | 37.0 (7.8)
    Siblings: number analyzed (Participants) | 52 | 54 | 106
    Siblings | 27.4 (7.9) | 24.4 (5.6) | 25.9 (7.0)
Child percent over median body mass index [Median (Full Range); unit: percent] — Body Mass Index (BMI) - BMI 50th percentile/BMI 50th percentile) × 100 Population: Percent over the age- and sex-specific 50th BMI percentile for kids, percent over the sex-specific 50th BMI percentile for 20-year-olds for parents. Parents are not included in this measurement. This measurement is to describe child body composition and not used for parents.
  percent
    Targeted Children: number analyzed (Participants) | 226 | 226 | 452
    Targeted Children | 53.8 [15.6 to 177.9] | 56.1 [15.9 to 187.2] | 54.7 [15.6 to 187.2]
    Sibling: number analyzed (Participants) | 52 | 54 | 106
    Sibling | 51.8 [12.2 to 200.7] | 37.3 [12.2 to 111.7] | 41.9 [12.2 to 200.7]
Child BMI percentile [Median (Full Range); unit: percentile] — Population: Parents are not included in this measurement. This measurement is to describe child body composition and not used for parents
  percentile
    Targeted Children: number analyzed (Participants) | 226 | 226 | 452
    Targeted Children | 98.46 [82.30 to 99.88] | 98.27 [83.56 to 99.81] | 98.40 [82.30 to 99.88]
    Siblings: number analyzed (Participants) | 52 | 54 | 106
    Siblings | 98.04 [87.12 to 100.0] | 96.96 [85.22 to 99.95] | 97.43 [85.22 to 100.00]

OUTCOME MEASURES:

1. Primary Outcome: Body Composition Measures of Targeted Child. Percent Change Over the Median BMI
Description: Height and weight will be taken to calculate changes in over weight status for children in FBT versus UC. Change in percent over median BMI from baseline to 24-month. Percent over the age- and sex-specific 50th BMI percentile for kids, percent over the sex-specific 50th BMI percentile for 20-year-olds for parents. Parents are not included in this measurement. This measurement is to describe child body composition and not used for parents. Results are pooled across 10 multiple imputations and reported as mean (standard error)
Time Frame: 0 - 24 months
Population: Targeted Children
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Usual Care (UC) | Family-based Treatment (FBT)
Number analyzed (Participants) | 226 | 226
percent change | 10.2 (1.0) | 3.4 (1.3)
Statistical Analysis 1: Comparison: Usual Care (UC) vs Family-based Treatment (FBT); Test type: Superiority; p < 0.05, ANCOVA; Mean Difference (Final Values) = -6.21, 95% CI 2-sided [-10.14 to -2.29] — Results are pooled across 10 multiple imputations and reported as mean (standard error)

2. Secondary Outcome: Body Composition Measures of Participating Parent. BMI (kg/m^2) Change From Baseline to 24 Month
Description: Height and weight will be taken to calculate changes in over weight status for parents in FBT versus UC. Results are pooled across 10 multiple imputations and reported as mean (standard error)
Time Frame: 0-24 months
Population: Participating Parents
Measure: Mean (Standard Deviation); unit: Change in kg/m^2 (BMI)
Arm/Group | Usual Care (UC) | Family-based Treatment (FBT)
Number analyzed (Participants) | 226 | 226
Change in kg/m^2 (BMI) | -0.03 (0.22) | -0.62 (0.24)
Statistical Analysis 1: Comparison: Usual Care (UC) vs Family-based Treatment (FBT); Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Final Values) = -3.97, 95% CI 2-sided [-5.68 to -2.26] — Results are pooled across 10 multiple imputations and reported as mean (standard error)

3. Secondary Outcome: Body Composition Measures, Siblings
Description: Height and weight will be taken for non-targeted siblings to determine if weight loss effects of FBT extend beyond the participating parent and child.
Time Frame: 0-24 months
Population: Siblings
Measure: Mean (Standard Deviation); unit: Change in % over median BMI
Arm/Group | Usual Care (UC) | Family-based Treatment (FBT)
Number analyzed (Participants) | 52 | 54
Change in % over median BMI | 8.3 (2.6) | 6.6 (2.9)

4. Secondary Outcome: Delay Discounting
Description: Delay discounting will be measured using an adjusting amount discounting task with a delayed reward of $100. K-values will be calculated and log-versions will be used due to skewness of k-values. More negative k-values indicate more delayed choices, which is considered better decision making
Time Frame: 0, and 24 months
Population: Parents and children are reported separately. Intent to treat was not used, number analyzed included parents and children with complete data (baseline and 24 month delay discounting measures). Siblings are not analyzed here.
Measure: Mean (Standard Deviation); unit: natural log
Arm/Group | Usual Care (UC) | Family-based Treatment (FBT)
Number analyzed (Participants) | 287 | 271
natural log
  Parent baseline delay discounting log k-value: number analyzed (Participants) | 158 | 146
  Parent baseline delay discounting log k-value | -5.98 (3.21) | -6.14 (2.54)
  Parent 24-month Delay discounting log k-value: number analyzed (Participants) | 158 | 146
  Parent 24-month Delay discounting log k-value | -6.45 (2.58) | -6.75 (2.43)
  Child baseline delay discounting log k-value: number analyzed (Participants) | 129 | 125
  Child baseline delay discounting log k-value | -4.37 (4.02) | -4.22 (3.48)
  Child 24-month Delay discounting log k-value: number analyzed (Participants) | 129 | 125
  Child 24-month Delay discounting log k-value | -4.76 (3.23) | -4.71 (2.62)
Statistical Analysis 1: Comparison: Usual Care (UC) vs Family-based Treatment (FBT); repeated measures analysis of variance for parent delay discounting changes from 0 to 24-month. This includes only parents with complete data for both time points and does not exclude based on johnson-bickel rules. Reporting time x group analysis; Test type: Superiority; p = 0.65, ANOVA; time x group analysis; Mean Difference (Final Values) = -0.5384
Statistical Analysis 2: Comparison: Usual Care (UC) vs Family-based Treatment (FBT); repeated measures analysis of variance for child delay discounting changes from 0 to 24-month. This includes only parents with complete data for both time points and does not exclude based on johnson-bickel rules. Reporting time x group analysis; Test type: Superiority; p = 0.87, ANOVA — time x group analysis; Mean Difference (Net) = -0.3913

ADVERSE EVENTS:
Time Frame: Adverse events and Serious Adverse events were collect over the full two year study, 24 month +/- 3 months.
Description: A systematic survey was administered at each measurement time point for the family. Non-systematic adverse events were collected by the coaches if they shared during treatment session with their coaches over the two year study.
Arm/Group | Usual Care (UC) | Family-based Treatment (FBT)
All-Cause Mortality (participants affected / at risk) | 0/504 | 0/506
Serious Adverse Events (participants affected / at risk) | 24/504 | 39/506
Other Adverse Events (participants affected / at risk) | 314/504 | 345/506
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Usual Care (UC) (N=504) | Family-based Treatment (FBT) (N=506)
Parent Doctor Visit (General disorders) | 0/226 (0) | 0/226 (0)
Parent Mental Health (Psychiatric disorders) | 2/226 (2) | 1/226 (1)
Parent Hospitalization (General disorders) | 11/226 (16) | 22/226 (26)
Parent Injury (General disorders) | 1/226 (1) | 0/226 (0)
Parent Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3/226 (3) | 1/226 (1)
Targeted Child Doctor Visit (General disorders) | 0/226 (0) | 1/226 (1)
Targeted Child Mental Health (Psychiatric disorders) | 5/226 (5) | 8/226 (9)
Targeted Child Hospitalizations (General disorders) | 1/226 (2) | 1/226 (1)
Targeted Child Injury (General disorders) | 0/226 (0) | 0/226 (0)
Sibling mental health (Psychiatric disorders) | 0/52 (0) | 3/54 (4)
Sibling hospitalization (General disorders) | 1/52 (1) | 2/54 (2)
Sibling Doctor Visit (General disorders) | 0/52 (0) | 0/54 (0)
Sibling Injury (General disorders) | 0/52 (0) | 0/54 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Usual Care (UC) (N=504) | Family-based Treatment (FBT) (N=506)
Parent Doctor appointments (General disorders) | 46/226 (73) | 68/226 (98) — Doctor visit
Parent Common Pediatric Event (General disorders) | 37/226 (42) | 28/226 (42) — Common Pediatric events include children and parents events that usually happen such as infections, rashes, aches and pains
Parent Mental Health (Psychiatric disorders) | 43/226 (54) | 49/226 (65)
Parent Injury (General disorders) | 34/226 (40) | 35/226 (43)
Targeted Child Doctor appointments (General disorders) | 27/226 (30) | 28/226 (30)
Targeted Child Common Pediatric Events (General disorders) | 50/226 (72) | 42/226 (69)
Targeted Child Mental Health (Psychiatric disorders) | 52/226 (73) | 48/226 (72)
Targeted Child Injury (General disorders) | 25/226 (28) | 47/226 (62)
Sibling Doctor Appointments (General disorders) | 9/52 (11) | 9/54 (9)
Sibling Common Pediatric Events (General disorders) | 17/52 (20) | 20/54 (31)
Sibling Mental Health (General disorders) | 7/52 (9) | 10/54 (19)
Sibling Injury (General disorders) | 8/52 (9) | 7/54 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT02873715/Prot_SAP_ICF_000.pdf